CLINICAL TRIAL: NCT04799275
Title: A Phase II/III Randomized Study of R-MiniCHOP With or Without CC-486 (Oral Azacitidine) in Participants Age 75 Years or Older With Newly Diagnosed Diffuse Large B Cell Lymphoma, Grade IIIB Follicular Lymphoma, Transformed Lymphoma, and High-Grade B-Cell Lymphomas With MYC AND BCL2 and/or BCL6 Rearrangements
Brief Title: Testing CC-486 (Oral Azacitidine) Plus the Standard Drug Therapy in Patients 75 Years or Older With Newly Diagnosed Diffuse Large B Cell Lymphoma
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: End of Initial Phase of Multi-phase protocol
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-01256; NCI-2020-01256 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1918 (Other: SWOG); S1918 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2021-03-13; First posted 2021-03-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Ann Arbor Stage III Diffuse Large B-Cell Lymphoma; Ann Arbor Stage IIX (Bulky) Diffuse Large B-Cell Lymphoma; Ann Arbor Stage IV Diffuse Large B-Cell Lymphoma; Diffuse Large B-Cell Lymphoma Activated B-Cell Type; Diffuse Large B-Cell Lymphoma Associated With Chronic Inflammation; Diffuse Large B-Cell Lymphoma Germinal Center B-Cell Type; Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; EBV-Positive Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Grade 3b Follicular Lymphoma; HHV8-Positive Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; High Grade B-Cell Lymphoma With MYC and BCL2 and/or BCL6 Rearrangements; High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; High Grade B-Cell Lymphoma, Not Otherwise Specified; Intravascular Large B-Cell Lymphoma; Lymphoplasmacytic Lymphoma; Nodular Lymphocyte Predominant B-Cell Lymphoma; Primary Cutaneous Diffuse Large B-Cell Lymphoma, Leg Type; T-Cell/Histiocyte-Rich Large B-Cell Lymphoma; Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Transformed Marginal Zone Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell, Marginal Zone | interventions — Specimen Handling; Cyclophosphamide; Doxorubicin; Azacitidine; cc-486; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (oral azacitidine, R-miniCHOP) (Experimental): Patients receive CC-486 PO for 7 days prior to cycle 1. Patients then receive CC-486 PO on days 8-21. Treatment repeats every 21 days for cycles 1-5 in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV (or SC for cycles 2-6), cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 1, and prednisone PO on days 1-5. Treatment repeats every 21 days for cycles 1-6 (6 cycles total) in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Oral Azacitidine; Drug: Prednisone; Other: Questionnaire Administration; Biological: Rituximab; Drug: Vincristine Sulfate
- Arm II (R-miniCHOP) (Active Comparator): Patients receive rituximab IV (or SC for cycles 2-6), cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 1, and prednisone PO on days 1-5. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Prednisone; Other: Questionnaire Administration; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Drug: Oral Azacitidine — Given PO
  Other Names: Azacitidine Oral; CC 486; CC-486; CC486; Onureg
  Arms: Arm I (oral azacitidine, R-miniCHOP)
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Other: Questionnaire Administration — Ancillary studies
Biological: Rituximab — Given IV or SC
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II/III trial compares the side effects and activity of oral azacitidine in combination with the standard drug therapy (reduced dose rituximab-cyclophosphamide, doxorubicin, vincristine, and prednisone [R-miniCHOP]) versus R-miniCHOP alone in treating patients 75 years or older with newly diagnosed diffuse large B cell lymphoma. R-miniCHOP includes a monoclonal antibody (a type of protein), called rituximab, which attaches to the lymphoma cells and may help the immune system kill these cells. R-miniCHOP also includes prednisone which is an anti-inflammatory medication and a combination of 3 chemotherapy drugs, cyclophosphamide, doxorubicin, and vincristine. These 3 chemotherapy drugs, as well as oral azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Combining oral azacitidine with R-miniCHOP may shrink the cancer or extend the time without disease symptoms coming back or extend patient's survival when compared to R-miniCHOP alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the addition of CC-486 (oral azacitidine) to R-miniCHOP results in excess toxicity compared to R-miniCHOP alone that would preclude the combination from being studied further. (Safety run-in) II. To determine if the CC-486 + R-miniCHOP regimen should be tested further (Phase III) against the control R-miniCHOP alone based on progression-free survival (PFS). (Phase II component) III. To compare the overall survival (OS) between CC-486 + R-miniCHOP and R-miniCHOP alone. (Phase III component)

SECONDARY OBJECTIVES:

I. To assess the feasibility of delivering at least 4 cycles of CC-486 with R-miniCHOP in this population.

II. To assess toxicity for CC-486 + R-miniCHOP and for R-miniCHOP. III. To compare complete response rates, as defined by Lugano 2014 classification, between CC-486 + R-miniCHOP and R-miniCHOP alone.

INTEGRATED CORRELATIVE GERIATRIC ASSESSMENTS:

I. To compare functioning as assessed by the S1918 Comprehensive Geriatric Assessment (S1918 CGA) between participants treated with CC-486 + R-miniCHOP versus R-miniCHOP alone.

II. To evaluate if frailty status (fit/unfit versus [vs] frail/superfrail) as assessed by the FIL tool is associated with OS.

III. To evaluate if frailty as measured by the FIL tool correlates with the summary frailty index as measured using components of the S1918 CGA.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE:

Beginning 7 days prior to starting [protocol treatment, all patients receive vincristine sulfate intravenously (IV) on day 1, and prednisone orally (PO) daily on days 1-7.

Patients are then randomized to 1 of 2 arms.

ARM I: Patients receive CC-486 PO for 7 days prior to cycle 1. Patients then receive CC-486 PO on days 8-21. Treatment repeats every 21 days for cycles 1-5 in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV (or subcutaneously [SC] for cycles 2-6), cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 1, and prednisone PO on days 1-5. Treatment repeats every 21 days for cycles 1-6 (6 cycles total) in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study.

ARM II: Patients receive rituximab IV (or SC for cycles 2-6), cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 1, and prednisone PO on days 1-5. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up periodically until 5 years from the date of registration.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed diffuse large B-cell lymphoma (DLBCL), Ann Arbor Stage IIX (bulky), III or IV. Participants with DLBCL transformed from follicular lymphoma (FL) or marginal zone lymphoma (MZL, including mucosa-associated lymphoid tissue [MALT] lymphomas), lymphoplasmacytic lymphoma (LPL), or nodular lymphocyte-predominant Hodgkin Lymphoma (NLPHL) are eligible. Participants with Grade IIIB follicular lymphoma (FL) or high-grade B-cell lymphomas with MYC and BCL2 and/or BCL6 rearrangements are also eligible. Participants with DLBCL that arose from prior CLL (Richter's transformation) are not eligible.
* As defined by the World Health Organization (WHO), eligible lymphoma subtypes include the following:

  * DLBCL, not otherwise specified (NOS)
  * DLBCL, germinal-center B-cell type (GCB)
  * DLBCL, activated B-cell type (ABC)
  * T-cell histiocyte-rich B-cell lymphomas (THRBCL)
  * Primary cutaneous DLBCL, leg type
  * Intravascular large B cell lymphoma
  * EBV+ DLBCL, NOS
  * DLBCL associated with chronic inflammation
  * HHV8+ DLBCL, NOS
  * High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements
  * High grade B-cell lymphoma, NOS
  * Follicular lymphoma grade 3b
* Participants must have staging imaging performed within 28 days prior to registration, as follows. Positron emission tomography (PET)-computed tomography (CT) baseline scans are strongly preferred; diagnostic quality magnetic resonance imaging (MRI), contrast-enhanced CT, or contrast-enhanced MRI scans are also acceptable if PET-CT is not feasible at baseline. Note: PET-CT will be required at end of treatment (EOT) and progression for response assessment. Participants must have measurable disease (at least one lesion with longest diameter ≥ 1.5 cm). All measurable lesions (longest diameter >= 1.5 cm) must be assessed within 28 days prior to registration. Tests to assess non-measurable disease must be performed within 42 days prior to registration.
* Participants with known human immunodeficiency virus (HIV)-infection are eligible providing they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test (must be within 26 weeks prior to registration). Participants with known HIV must have a CD4 count checked within 28 days prior to registration, but may proceed with therapy regardless of CD4 count.
* All participants must be screened for chronic hepatitis B virus (HBV) within 28 days prior to registration. Participants with known HBV infection (positive serology) must also have a HBV viral load performed within 28 days prior to registration, and participants must have an undetectable HBV viral load on suppressive therapy within 28 days prior to registration. Participants found to be HBV carriers during screening are eligible and must receive standard of care prophylaxis. Participants with active hepatitis B (HBV viral load > 500 IU/mL) within 28 days prior to registration are not eligible
* Participants with a known history of hepatitis C virus (HCV) infection must have an undetectable HCV viral load within in 28 days prior to registration
* Participants must not have known lymphomatous involvement of the central nervous system (CNS)
* Participants must not have active inflammatory bowel disease (such as, Crohn's disease, ulcerative colitis), celiac disease (i.e., sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism, or excretion of the study drug and/or predispose the subject to an increased risk of gastrointestinal toxicity
* Participants must not have a history of acute leukemia having been treated with intensive induction therapy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Participants must not have received any prior cytotoxic chemotherapy or rituximab for treatment of the newly diagnosed DLBCL except for the pre-phase treatment (within specified dose range) that may have either started before or may start after registration to S1918. Inhaled, nasal, and topical steroid use is allowed. Prior cytotoxic chemotherapy and/or antibody therapy for an indolent lymphoma prior to transformation is allowed. Up to 4 doses of intrathecal (IT) chemotherapy administered for central nervous system (CNS) prophylaxis is allowed in addition to protocol therapy. High-dose intravenous methotrexate is not allowed.
* Participants must not have received more than a cumulative of dose 250 mg/m^2 of prior doxorubicin (or equivalent dose of another anthracycline, such as epirubicin) therapy (at any time prior to registration).
* Participants must not currently be receiving any other investigational agents
* Participant must not have a history of allergic reactions attributed to azacitidine, mannitol, or other hypomethylating agents
* Participants must be age ≥ 75
* Participants must have a Zubrod performance status of 0-2
* Participants must have adequate renal function, as demonstrated by a creatinine clearance, calculated by the Cockcroft and Gault formula, of >= 30 ml/min that was obtained within 28 days prior to registration
* Aspartate aminotransferase (AST) =< 2.5 x institutional upper limit of normal (IULN), alanine aminotransferase (ALT) =< 2.5 x IULN (within 28 days prior to registration)
* Total bilirubin =< 2 x institutional upper limit of normal (IULN), unless due to Gilbert's disease, hemolysis, or lymphomatous involvement of liver (within 28 days prior to registration). Note: If total bilirubin is elevated, and direct bilirubin is subsequently performed (within 28 days prior to registration) and resulted to be =< 2 x IULN, the participant will be considered eligible
* Absolute neutrophil count (ANC) >= 1000/mcL (within 28 days prior to registration)
* Platelets >= 75,000/mcL (within 28 days prior to registration)
* Hemoglobin (Hgb) >= 8 g/ dL (within 28 days prior to registration)
* If there is a documented lymphomatous involvement of the bone marrow, bone marrow function within 28 days prior to registration, as evidenced by:

  * ANC >= 500/mcL
  * Platelets >= 50,000/mcL
  * Hemoglobin (Hgb) >= 8 g/ dL
* Participants must have a left ventricular ejection (LVEF) fraction >= 45% as measured by echocardiogram or radionuclide (multigated acquisition scan [MUGA]) ventriculography within 56 days prior to registration
* For the duration of the study treatment period and for at least 4 months following the last dose of study drug, male participants must agree to use effective contraceptive methods during sexual contact with a female of childbearing potential (FCBP) and must agree to refrain from semen or sperm donation during the same timeframe. Effective contraceptive methods include a history of vasectomy, use of hormonal contraception or an intrauterine device (IUD) by the female partner, or use of condoms

  * A FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Participants must not have active infection (systemic fungal, bacterial, or viral infection) that is not controlled (defined as ongoing signs/symptoms related the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
* Participants must not have active cardiac disease within 26 weeks prior to registration, including: symptomatic congestive heart failure (New York Heart Association [NYHA] class 4), unstable angina pectoris, hemodynamically unstable cardiac arrhythmia, or myocardial infarction
* Participants must not have >= grade 2 neuropathy, by Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 5.0, within 28 days prior to registration
* Participants must not have any other known uncontrolled intercurrent illness including, but not limited to ongoing psychiatric illness/social situations that would limit compliance with study requirements
* Participants must not have a concurrent primary malignancy undergoing active therapy. Exceptions: participants may have non-melanomatous skin cancers requiring only surgical intervention. Participants may have a history of early stage breast cancer or prostate cancer in remission after surgical and/or radiation therapy on adjuvant hormonal therapy only

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Excess toxicity as a result of adding oral azacitidine (CC-486) to reduced dose rituximab-cyclophosphamide, doxorubicin, vincristine, and prednisone (R-miniCHOP) (Safety run-in) | Up to completion of cycle 6
  Will determine if the addition of CC-486 to R-miniCHOP results in excess toxicity compared to R-miniCHOP alone that would preclude the combination from being studied further.
Progression-free survival (PFS) (Phase II) | From date of registration to date of first observation of progressive disease according to the 2014 Lugano classification, or death due to any cause, assessed up to 1 year
  Will determine if the CC-486 + R-miniCHOP regimen should be tested further (Phase III) against the control R-miniCHOP alone based on PFS. After accruing 130 patients (65 per arm, 21 months of accrual and potentially pausing accrual for 6 months follow-up to reach a target 63 events across arms), a one-sided stratified .10 log-rank test will inform a go/no-go decision based on sufficient evidence of efficacy to continue to the Phase III portion of the study.
Overall survival (Phase III) | From date of registration to date of death due to any cause, assessed up to 2 years
  Will compare overall survival in the control arm of R-miniCHOP to the experimental arm of CC-486 (oral azacitidine) + R-miniCHOP. Will be evaluated using a 1-sided .025 level stratified logrank test.

SECONDARY OUTCOMES:
Metabolic complete response (CR) | Up to end of cycle 6 or end of treatment
  Will be defined using 2014 Lugano classification. Fisher's exact test will be used to compare CR rates between the experimental arm of CC-486 + R-miniCHOP and the control arm of R-miniCHOP alone.
Incidence of adverse events | Until disease progression, assessed up to 5 years
  Will be assessed using Common Terminology Criteria for Adverse Events version 5. The maximum Grade for each toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. Treatment-related toxicities between arms will be compared using Fisher's exact test.
Overall survival (Phase III) | From date of registration to date of death due to any cause, assessed up to 5 years
  An additional secondary analysis of overall survival of the Phase III comparison will adjust for patients with identified double-hit phenotype in addition to the pre-specified stratification factors. Will also prospectively collect the number of days between diagnostic biopsy and cycle 1 day 1 of therapy for a pre-planned secondary analysis.

OTHER OUTCOMES:
Changes in function (Integrated Correlative Geriatric Assessments Substudy) | From time of randomization up to 24 months after date of registration
  Will be assessed by a Comprehensive Geriatric Assessment (Carolina Frailty Index [CFI] Score) between patients treated with CC-486 + R-miniCHOP and those treated with R-miniCHOP alone. Linear regression will be used for each examination, adjusting for the stratification factors from the clinical study and the baseline score (for the examination of change from 12 to 24 months, the 12-month score will be considered the baseline score). Although the number of timepoints is limited to 3, longitudinal assessments of the CFI Score over time will also be conducted using linear mixed models, adjusting for the stratification factors and the baseline score, with patient considered a random effect.
Frailty status (fit/unfit vs frail) (Integrated Correlative Geriatric Assessments Substudy) | Baseline
  Will evaluate if frailty status (fit/unfit versus frail) as assessed by the Italian Lymphoma Foundation (FIL) tool is associated with overall survival. Multivariable Cox regression will be conducted, adjusting for the stratification variables and the randomized treatment arm as covariates. Will also examine whether randomization to CC-486 + R-miniCHOP is associated with better overall survival compared to treatment with R-miniCHOP alone in the subset of fit and unfit patients. Multivariable Cox regression will be conducted, adjusting for the stratification variables as covariates.
Frailty status (Integrated Correlative Geriatric Assessments Substudy) | Up to 24 months after date of registration
  Will evaluate if frailty status (fit/unfit versus frail) as assessed by the FIL tool correlates with the summary frailty indexed as measured by the S1918 Comprehensive Geriatric Assessment (CGA). In particular, agreement between the FIL and CGA will measured using an unweighted Kappa statistic; moderate or better agreement is defined as a Kappa coefficient of >= 0.41.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Brem, Principal Investigator — SWOG Cancer Research Network
Locations (176):
- United States (176):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente South Bay, Harbor City, California
  - City of Hope Seacliff, Huntington Beach, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Kaiser Permanente-Irvine, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - City of Hope Newport Beach, Newport Beach, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - UCSF Cancer Center - San Mateo, San Mateo, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope South Bay, Torrance, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Lutheran Hospital - Cancer Centers of Colorado, Golden, Colorado
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - George E Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - FHCC Overlake, Bellevue, Washington
  - FHCC at EvergreenHealth, Kirkland, Washington
  - FHCC at Northwest Hospital, Seattle, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Brem EA, Li H, Beaven AW, Caimi PF, Cerchietti L, Alizadeh AA, Olin R, Henry NL, Dillon H, Little RF, Laubach C, LeBlanc M, Friedberg JW, Smith SM. SWOG 1918: A phase II/III randomized study of R-miniCHOP with or without oral azacitidine (CC-486) in participants age 75 years or older with newly diagnosed aggressive non-Hodgkin lymphomas - Aiming to improve therapy, outcomes, and validate a prospective frailty tool. J Geriatr Oncol. 2022 Mar;13(2):258-264. doi: 10.1016/j.jgo.2021.10.003. Epub 2021 Oct 20. PMID 34686472